CLINICAL TRIAL: NCT05975632
Title: GAMMA Study: Patient Self-testing of Capillary Blood Potassium: A Validation Study and Measurement Performance in Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CardioRenal (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR-2023-001
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Potassium Measurement
Keywords: self-test; capillary collection; in-vitro diagnostic medical device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Potassium measurement (Experimental): Calibration Phase : 1 visit (duration 1 day) for subjects not on dialysis and hemodialysis patients Comparaison Phase : 1 visit (diration 1 day) for hemodialysis patients Comparaison Phase : 2 visits (diration 1 day) for subjects not on dialysis
  Interventions: Device: Device: Self testing Potassium device

INTERVENTIONS:
Device: Device: Self testing Potassium device — Calibration Phase (1 visit) (Hemodialysis patients and subjects not on dialysis) Each patient will have one venous blood collection. Among them, one 30 patients one capillary sample is collected. In this phase, the HCP is the user of the device.
  Comparison Phase
  For subject not on dialysis (total 2 visits):
  Each patient will have one venous blood collection per visit Each patient will be equipped with CardioRenal device and trained to do the self-test
  For Hemodialysis patients (total 1 visit) :
  Each patient will have one venous blood collection per visit Each patient will be equipped with CardioRenal device and trained to do the self-test

SUMMARY:
Multicentre, open, prospective and interventional study investigating the CardioRenal device in capillary blood of patients.It will be conducted at multiple investigational sites.

DETAILED DESCRIPTION:
Objectives are to assess the quantitative accuracy in freshly collected whole capillary blood from patients and healthy volunteers and to evaluate user proficiency. In order to gather a wide range of K+ concentrations, the study will be conducted both on patients or healthy volunteers and on dialysis patients.

The study includes 2 phases (calibration phase and comparison phase) where blood samples (capillary and venous) will be collected.Blood is taken from the subject by trained specialist staff. During the comparison phase, the subjects will be equipped with CardioRenal device and trained to do the self-test.

A subject's participation in this study (both calibration and validation phase) will consist of two interventional visits for hemodialysis patients and three interventional visits for other subjects.

ELIGIBILITY:
Inclusion Criteria for subjects not on dialysis:

* Male/female subject, aged 18+ years ;
* Signing a written informed consent ;
* Willing to perform the self-test after viewing the instruction for use;
* Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Inclusion Criteria for hemodialysis patients:

* Male/female subject, aged 18+ years ;
* Medical history of dyskalemia ;
* Signing a written informed consent ;
* Willing to perform the self-test after viewing the instruction for use;
* Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Non-inclusion Criteria for subjects not on dialysis:

* Medical history of seizure (epilepsy)
* Known inherited hemolytic anemia
* Autoimmune hemolytic anemia
* Infectious Hemolytic anemia
* Prosthetic Cardiac valves
* Hemolytic uremic syndrome
* Peripheral edema
* Dehydration
* Peripheral Arterial Obstructive Disease (PAOD) stage 4
* Raynaud syndrome
* Known evolutive cancers
* Subjects who are pregnant or breast-feeding
* Vulnerable patients, patients deprived from liberty and patients with a physical or mental state altered by disease, age or disability which impacts their ability to defend their interests and for which protection measures are taken
* Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development
* Subject who is prohibited from participation in the study after consulting the Ministry of Health National File (e.g. indemnities > 6000 euros for a 12-months period)

Non-inclusion Criteria for hemodialysis patients:

* Medical history of seizure (epilepsy)
* Known inherited hemolytic anemia
* Autoimmune hemolytic anemia
* Infectious Hemolytic anemia
* Prosthetic Cardiac valves
* Hemolytic uremic syndrome
* Peripheral edema
* Dehydration
* Peripheral Arterial Obstructive Disease (PAOD) stage 4
* Raynaud syndrome
* Known evolutive cancers
* Subjects who are pregnant or breast-feeding
* Vulnerable patients, patients deprived from liberty and patients with a physical or mental state altered by disease, age or disability which impacts their ability to defend their interests and for which protection measures are taken
* Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development
* Subject who is prohibited from participation in the study after consulting the Ministry of Health National File (e.g. indemnities > 6000 euros for a 12-months period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Calibrations factors and correlations R² | through study completion, an average of 3 months
  potassium values
Accuracy of measurement of the capillary whole blood potassium with TENOR compared to the reference method (indirect potentiometry) | through study completion, an average of 3 months
  potassium values

SECONDARY OUTCOMES:
Determination of mean, standard deviation (SD) and coefficient of variation (CV) | through study completion, an average of 3 months
  repeatability
Usability Evaluation questionnaire | through study completion, an average of 3 months

OTHER OUTCOMES:
Record and evaluate adverse events | through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Louis Carron, MD, Principal Investigator — CHU Grenoble-Alpes Service de Nephrologie
Locations (6):
- France (6):
  - Centre d'Investigation Clinique, Grenoble
  - CHU Grenoble-Alpes, Grenoble
  - Agduc La Tronche, La Tronche
  - Diaverum, Marseille
  - Hôpital Saint Joseph, Marseille
  - Biogroup, Meylan